CLINICAL TRIAL: NCT07027761
Title: Maternal Mental Health Intervention (MaMHI) Study: A Combined Non-inferiority and Superiority Randomized Controlled Trial Comparing the Clinical and Cost-effectiveness of an Online Self-help Intervention and a Brief Face-to-face Intervention Versus Usual Care in Mothers at Moderate Risk for Perinatal Depression Identified by a Concentration-of-risk Prediction Approach.
Brief Title: Clinical and Cost-effectiveness of an Online Self-help Intervention and a Face-to-face Intervention Versus Usual Care in Mothers at Moderate Risk for Perinatal Depression
Acronym: MaMHI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Erasmus University Rotterdam (Other)
Responsible Party: Principal Investigator, PATRICK LUYTEN, Full Professor of Clinical Psychology, KU Leuven, Belgium, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S64351; C24M/22/054 (Other: KU Leuven)
Record Dates: First submitted 2025-06-02; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Perinatal Depression
Keywords: Perinatal depression; maternal mental health; face-to-face intervention; online self-help; early intervention, brief psychotherapy; psychodynamic therapy.

STUDY DESIGN:
Intervention Model Description: A single-site, assessor-blinded, combined superiority and non-inferiority randomized controlled trial comparing an online self-help intervention (+ usual care) and a brief face-to-face intervention (+ usual care) with usual care in mothers at moderate risk for perinatal depression.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online self-help (Active Comparator): Online Self-Help refers to a 24/7 accessible, internet-based platform that offers digital modules grounded in evidence-based approaches, including infant mental health, cognitive-behavioral therapy (CBT), and psychodynamic interventions, aimed at addressing perinatal depression (https://perinatalehulp.be/).
  Interventions: Behavioral: Online self-help
- Maternal Mental Health Intervention (MaMHI) (Active Comparator): A brief, eight-session face-to-face intervention designed for (expectant) mothers and their infants across the perinatal period.
  Interventions: Behavioral: Maternal Mental Health Intervention (MaMHI)
- Usual care (Other): Usual care offered to (expectant) mothers in Flanders, Belgium
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Online self-help — Online Self-Help refers to a 24/7 accessible, internet-based platform that offers digital modules grounded in evidence-based approaches, including infant mental health, cognitive-behavioral therapy (CBT), and psychodynamic interventions, aimed at addressing perinatal depression (https://perinatalehulp.be/). Upon logging in, participants receive an overview of the available modules and can select from three distinct treatment trajectories, ideally to be completed over the course of 10 weeks: (a) a self-directed option allowing free choice among all modules; (b) a structured CBT trajectory incorporating both second-wave and third-wave cognitive-behavioral strategies; or (c) a psychodynamic trajectory primarily focused on relational and attachment-related factors contributing to the onset and maintenance of perinatal depression.
  Arms: Online self-help
Behavioral: Maternal Mental Health Intervention (MaMHI) — A brief, eight-session face-to-face intervention designed for (expectant) mothers and their infants across the perinatal period, consisting of four prenatal sessions (during the second and third trimesters of pregnancy) and four postnatal sessions conducted within the first three months postpartum. The intervention is grounded in psychodynamic principles and informed by mentalization-based approaches
  Arms: Maternal Mental Health Intervention (MaMHI)
Other: Usual Care — Prenatal care is provided through follow-up by a general practitioner and a gynecologist and/or a midwife, while postnatal follow-up is conducted by Child and Family Care Services.
  Arms: Usual care

SUMMARY:
The perinatal period (pregnancy and the first postnatal year) (O'Hara & Wisner, 2014) involves important changes and considerable challenges for parents (Milgrom & Gemmill, 2015). As a result, perinatal mental health (PMH) disorders are highly prevalent. It is estimated that 1 in 5 women meet criteria for mental health disorders during the perinatal period (Van Damme et al., 2018). These psychological problems not only significantly impact (expectant) mother's own wellbeing, but also that of their children, partners, and their support networks. Additionally, PMH problems are associated with significant financial burden. For instance, In the UK perinatal depression and anxiety are estimated to cost approximately £8.1 billion per annual birth cohort (Bauer, 2015). Prevention of these problems is therefore essential. Unfortunately, in up to 75% of women symptoms of depressive or anxiety disorders are not detected timely, and only 10% of these women receive appropriate help (Kingston et al., 2015).

This study proposes a novel approach to intervention by investigating the effectiveness of psychosocial treatments for (expectant) mothers identified to be at moderate risk of developing perinatal depression based on a novel statistical risk modeling approach. Specifically, we will investigate the clinical and cost-effectiveness of (a) an online self-help program and (b) a brief face-to-face (FTF) intervention for expectant mothers with a moderate risk of developing perinatal depression, compared to (c) standard care (treatment as usual). We expect both active treatments to be superior compared to standard care and similar in effectiveness to each other. In addition, we expect both online self-help and the brief FTF intervention to be more cost-effective compared to usual care. Moreover, we will also investigate the effects of the three treatments on a range of other important outcomes, participants' satisfaction with the treatments, the credibility of the treatments and expected effects as rated by patients. Finally, in a small qualitative study, we will investigate the subjective experiences of participants in the brief FTF intervention specifically.

DETAILED DESCRIPTION:
Introduction The perinatal period, encompassing pregnancy and the first year postpartum (O'Hara & Wisner, 2014), represents a time of significant physiological, psychological and social change, necessitating considerable adaptation by expectant parents (Milgrom & Gemmill, 2015). This transitional phase is characterized by a coexistence of intense positive emotions-such as joy, hope, and excitement-and challenging negative emotions, including insecurity, anxiety and depression. As a result, both the transition to parenthood and the early stages of parenting are associated with increased vulnerability to emotional difficulties.

Mental health problems are highly prevalent in the perinatal period, affecting approximately one in five expectant or new mothers (Van Damme et al., 2018). Among these, perinatal depression (PD)-which includes both minor and major depressive episodes-is one of the most common complications during pregnancy and postpartum (Wisner et al., 2013). The point prevalence of major depressive disorder during pregnancy ranges from 3.1% to 4.9%, increasing to approximately 5% in the first three months postpartum. Minor depression affects an estimated 11% of pregnant women and 13% of women in the first three months after childbirth. The period prevalence of any depression during pregnancy and the first three postpartum months is estimated at 18.4% and 19.2%, respectively, with 12.7% and 7.1% meeting criteria for major depression during those timeframes (Gavin et al., 2005). Notably, one-third of postpartum depression cases begin during pregnancy, and 27% have onset prior to pregnancy (Wisner et al., 2013). Depression during the second and third trimesters increases the likelihood of postpartum depression by factors of 3.2 and 6.6, respectively (Heron et al., 2004). Mental health disturbances during pregnancy are therefore strong predictors of postpartum mental health status (Robertson et al., 2004).

Although most women recover from postnatal depression within a few months, approximately 30% remain clinically depressed beyond the first postpartum year (Goodman, 2004), and 40% may develop a chronic depressive disorder (Vliegen et al., 2014).

The consequences of perinatal depression extend beyond the individual, significantly affecting the mother-infant relationship and the child's socio-emotional development (Atif et al., 2015). For instance, the perinatal period is critical for the establishment of a secure attachment, which is fundamental to a mother's capacity to recognize and respond to her infant's emotional cues (Rosenboom, 2018). Maternal mental health issues may interfere with mothers' emotional availability and responsiveness, which may in turn compromise children's development.

Consistent with these assumptions, epidemiological and longitudinal studies have demonstrated that children of parents with depression have significantly elevated risks of developing depression themselves (Rosenboom, 2018). For example, Weissman et al. (2006) found that offspring of depressed parents were three to four times more likely to develop depression compared to children of non-depressed parents, with up to 50% affected by age 20.

Perinatal mental health (PMH) problems are associated with a high socio-economic burden. According to a UK report by Bauer et al. (2015), the annual cost of PMH problems in the United Kingdom was estimated at £8.1 billion per birth cohort, with 72% of this cost attributed to adverse impacts on child development (Sutter-Dallay et al., 2016). Early identification and intervention are therefore critical for reducing both the prevalence and economic burden of PMH issues (Sutter-Dallay et al., 2016).

Despite robust evidence on the impact of PD and broader PMH disorders on maternal, infant and family well-being, early detection and prevention remain problematic. Approximately 75% of women experiencing perinatal anxiety or depression go undiagnosed, and only about 10% of expectant and new mothers receive adequate treatment (Kingston et al., 2015). In this context, brief and low-intensity interventions show promise, with meta-analytic evidence supporting the efficacy of brief (preventative) interventions, including digital formats (Loughnan et al., 2019).

However, access to these interventions is often restricted to individuals with subthreshold symptoms or those highly motivated to seek care. Interventions that match the risk status of individuals may be more effective than a 'one-size-fits-all' approach. For instance, for women with more complex and persistent depression, targeted intensive approaches may be most effective (Howard & Khalifeh, 2020). Women with less severe clinical presentations may respond well to brief, scalable interventions, including online self-help programs and brief face-to-face (FTF) psychological interventions (Loughnan et al., 2019), and these interventions may also be cost-effective.

The present study This study will be the first to evaluate the clinical and cost-effectiveness of an online self-help intervention compared to a brief 8-session FTF intervention, both offered alongside usual care, for pregnant women at moderate risk for developing PD based on an analytical epidemiological approach aligned with precision medicine principles relying on a concentration-of-risk prediction modeling approach.

The primary aim of this study is to assess whether an online self-help program and a brief FTF intervention, in conjunction with usual care, is superior to usual care alone in reducing severity of depression from baseline to end-of-treatment (primary outcome). It is hypothesized that both interventions will be superior to usual care and that online self-help is non-inferior to the brief FTF intervention.

Secondary aims are to assess whether online self-help and brief FTF intervention are more effective than usual care in reducing parental stress, and in fostering mother-infant bonding, child socio-emotional development, and quality of life (secondary outcomes).

In addition, treatment credibility and expectancy of and satisfaction with the three treatments will be investigated, as well as their cost-effectiveness.

A qualitative study will be embedded within the trial to investigate mothers' experience of the brief FTF intervention.

References

Atif, N., Lovell, K., & Rahman, A. (2015). Maternal mental health: The missing "m" in the global maternal and child health agenda. Seminars in Perinatology, 39, 345-352. https://doi.org/10.1053/j.semperi.2015.06.007 Bauer, A., Pawlby, S., Plant, D. T., King, D., Pariante, C. M., & Knapp, M. (2015). Perinatal depression and child development: exploring the economic consequences from a South London cohort. Psychological Medicine, 45(1), 51-61. https://doi.org/10.1017/S0033291714001044 Berry, J. O., & Jones, W. H. (1995). The Parental Stress Scale: Initial Psychometric Evidence. Journal of Social and Personal Relationships, 12(3), 463-472. https://doi.org/10.1177/0265407595123009 Bouwmans, C., De Jong, K., Timman, R., Zijlstra-Vlasveld, M., Van der Feltz-Cornelis, C., Tan, S. S., & Hakkaart-van Roijen, L. (2013). Feasibility, reliability and validity of a questionnaire on healthcare consumption and productivity loss in patients with a psychiatric disorder (TiC-P). BMC Health Services Research, 13(1), 217. https://doi.org/10.1186/1472-6963-13-217 Condon, J. T., & and Corkindale, C. J. (1998). The assessment of parent-to-infant attachment: Development of a self-report questionnaire instrument. Journal of Reproductive and Infant Psychology, 16(1), 57-76. https://doi.org/10.1080/02646839808404558 Cox, J. L., Holden, J. M., & Sagovsky, R. (1987). Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry, 150, 782-786. https://doi.org/10.1192/bjp.150.6.782 Devilly, G. J., & Borkovec, T. D. (2000). Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry, 31(2), 73-86. https://doi.org/10.1016/s0005-7916(00)00012-4 Feinberg, M. E., D., B. L., & and Kan, M. L. (2012). A Multi-Domain Self-Report Measure of Coparenting. Parenting, 12(1), 1-21. https://doi.org/10.1080/15295192.2012.638870 Gavin, N. I., Gaynes, B. N., Lohr, K. N., Meltzer-Brody, S., Gartlehner, G., & Swinson, T. (2005). Perinatal depression: a systematic review of prevalence and incidence. Obstet Gynecol, 106(5 Pt 1), 1071-1083. https://doi.org/10.1097/01.AOG.0000183597.31630.db Goodman, J. H. (2004). Postpartum Depression Beyond the Early Postpartum Period. Journal of Obstetric, Gynecologic & Neonatal Nursing, 33(4), 410-420. https://doi.org/https://doi.org/10.1177/0884217504266915 Herdman, M., Gudex, C., Lloyd, A., Janssen, M., Kind, P., Parkin, D., Bonsel, G., & Badia, X. (2011). Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res, 20(10), 1727-1736. https://doi.org/10.1007/s11136-011-9903-x Heron, J., O'Connor, T. G., Evans, J., Golding, J., & Glover, V. (2004). The course of anxiety and depression through pregnancy and the postpartum in a community sample. Journal of Affective Disorders, 80(1), 65-73. https://doi.org/https://doi.org/10.1016/j.jad.2003.08.004 Howard, L. M., & Khalifeh, H. (2020). Perinatal mental health: a review of progress and challenges. World Psychiatry, 19(3), 313-327.

Kingston, D., Austin, M.-P., Heaman, M., McDonald, S., Lasiuk, G., Sword, W., Giallo, R., Hegadoren, K., Vermeyden, L., van Zanten, S. V., Kingston, J., Jarema, K., & Biringer, A. (2015). Barriers and facilitators of mental health screening in pregnancy. Journal of Affective Disorders, 186, 350-357. https://doi.org/https://doi.org/10.1016/j.jad.2015.06.029 Loughnan, S. A., Joubert, A. E., Grierson, A., Andrews, G., & Newby, J. M. (2019). Internet-delivered psychological interventions for clinical anxiety and depression in perinatal women: a systematic review and meta-analysis. In (Vol. 22, pp. 737-750): Springer-Verlag Wien.

Milgrom, J., & Gemmill, A. W. (2015). Identifying Perinatal Depression and Anxiety: Evidence-Based Practice in Screening, Psychosocial Assessment, and Management. John Wiley & Sons. https://doi.org/10.1002/9781118509722 O'Hara, M. W., & Wisner, K. L. (2014). Perinatal mental illness: Definition, description and aetiology. Best Practice & Research Clinical Obstetrics & Gynaecology, 28(1), 3-12. https://doi.org/https://doi.org/10.1016/j.bpobgyn.2013.09.002 Robertson, E., Grace, S., Wallington, T., & Stewart, D. E. (2004). Antenatal risk factors for postpartum depression: a synthesis of recent literature. General Hospital Psychiatry, 26(4), 289-295. https://doi.org/https://doi.org/10.1016/j.genhosppsych.2004.02.006 Rosenboom, T. (2018). De eerste 1000 dagen: het fundamentele belang van een goed begin vanuit biologisch, medisch en maatschappelijk perspectief. de Tijdstroom.

Squires, J., Bricker, D., Twombly, E., Hoselton, R., Murphy, K., Dolata, J., Yockerlson, S., Schoen Davis, M., & Kim, Y. (2015). A Parent-Completed Child Monitoring System for Social-Emotional Behaviors Ages & Stages Questionnaires: Social-Emotional.

Sutter-Dallay, A.-L., Glangeaud-Freudenthal, N. M.-C., Guedeney, A., & Riecher-Rössler, A. (2016). Joint Care of Parents and Infants in Perinatal Psychiatry (1st ed.). Springer International Publishing Switzerland.

Van Damme, R., Van Parys, A.-S., Vogels, C., Roelens, K., & Lemmens, G. (2018). Screening en detectie van perinatale mentale stoornissen: richtlijn als leidraad voor het ontwikkelen van een zorgpad. UZ Gent; Universiteit Gent; Karus, Vlaanderen is zorg.

Vliegen, N., Casalin, S., & Luyten, P. (2014). The Course of Postpartum Depression: A Review of Longitudinal Studies. Harvard Review of Psychiatry, 22(1). https://journals.lww.com/hrpjournal/fulltext/2014/01000/the_course_of_postpartum_depression__a_review_of.1.aspx Weissman, M. M., Wickramaratne, P., Nomura, Y., Warner, V., Pilowsky, D., & Verdeli, H. (2006). Offspring of depressed parents: 20 years later. Am J Psychiatry, 163(6), 1001-1008. https://doi.org/10.1176/ajp.2006.163.6.1001 Wisner, K. L., Sit, D. K. Y., McShea, M. C., Rizzo, D. M., Zoretich, R. A., Hughes, C. L., Eng, H. F., Luther, J. F., Wisniewski, S. R., Costantino, M. L., Confer, A. L., Moses-Kolko, E. L., Famy, C. S., & Hanusa, B. H. (2013). Onset Timing, Thoughts of Self-harm, and Diagnoses in Postpartum Women With Screen-Positive Depression Findings. JAMA Psychiatry, 70(5), 490-498. https://doi.org/10.1001/jamapsychiatry.2013.87

ELIGIBILITY:
Inclusion Criteria:

Participants will be drawn from the broader PRIL (Perinatal mental health Profiling and Intervention in Leuven) study, who consented to being contacted for the intervention trial and who meet criteria for moderate risk for perinatal depression based on an analytical epidemiological approach aligned with precision medicine principles, specifically a concentration-of-risk prediction modeling approach. Based on a comprehensive assessment of biological, psychological and social risk and protective factors, concentration-of-risk models will be developed and validated to stratify respondents in terms of risk for future perinatal depression, namely (1) not, (2) mildly, (3) moderately and (4) highly at risk of developing perinatal depression. Mothers falling into the moderate risk profile are eligible to participate

Exclusion Criteria:

* Receiving concurrent psychological guidance in perinatal mental health problems;
* Not consenting to (a) audiorecording of the first two face-to-face sessions and/or (b) paying the appropriate fee, in case of randomization to the face-to-face intervention arm.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Changes in perinatal depressive symptoms, as measured by the Edinburgh (Postnatal) Depression Scale (E(P)DS), from baseline to end-of-treatment (EOT). | EOT (i.e., at 3 months postpartum)
  Severity of perinatal depression as measured by the E(P)DS (Cox et al., 1987)(range 0 - 30, with higher scores reflecting worse outcome).

SECONDARY OUTCOMES:
Changes in perinatal depressive symptoms, as measured by the Edinburgh (Postnatal) Depression Scale (E(P)DS), from baseline to 12-months follow-up | 12 months follow-up
  Severity of depression as measured by the EPDS (Cox et al., 1987). Scores range from 0 to 30, with higher scores reflecting higher levels of perinatal depression
Parental stress, as measured by the Parental Stress Scale (PSS), at EOT and 12-months follow-up; | EOT (i.e., at 3 months postpartum) and 12-months follow-up
  Parental stress as measured by the Parental Stress Scale (PSS; Berry & Jones, 1995). The PSS measures the levels of stress experienced by parents taking into account positive and negative aspects of parenting. Scores range between 18 and 90, with higher scores reflecting higher perceived parental stress
Changes in mother-infant bonding, as measured by the Maternal Postnatal Attachment Scale (MPAS), from baseline to EOT and 12-months follow-up | EOT (i.e., at 3 months postpartum) and 12-month follow-up
  Mother-infant bonding as measured by the Maternal Postnatal Attachment Scale (MPAS; Condon & and Corkindale, 1998). The MPAS measures the emotional tie or bond of a mother towards her infant through self-reported feelings, cognitions and behaviors. The scale comprises three subscales: quality of attachment, pleasure in interaction, and absence of hostility. Total scores range between 19 and 95, with higher scores indicating stronger mother-infant bonding. The subscale scores range from 9 to 45 for quality of attachment and 5 to 25 for both pleasure in interaction and absence of hostility
Child socio-emotional development, as measured by the Ages & Stages Questionnaire - Social-Emotional (ASQ:SE-2), at EOT and 12-months follow-up | EOT (i.e., at 3 months postpartum) and 12-months follow-up
  Child socio-emotional development as measured by the Ages & Stages Questionnaire - Social-Emotional (ASQ:SE-2; Squires et al., 2015). The ASQ:SE-2 assesses various dimensions of children's social-emotional development, screening for potential delays and identifying children at risk for developmental problems. The questionnaire is completed by the primary caregiver and can be administered to children aged 3 to 66 months, using the version closest to the child's age (available for 6, 12, 18, 24, 30, 36, 48, and 60 months). Parents indicate how often the child exhibits the described behavior: "most of the time" (0 points), "sometimes" (5 points), or "rarely/never" (10 points). Additionally, parents can express concerns about specific behaviors, adding 5 extra points per marked item. Given the age range of our sample, the 6- and 12-month versions are used. Total scores are calculated by summing all item points and expressed concerns, with higher scores indicating lower levels of child
Coparenting, as measured by the Coparenting Relationship Scale (CRS; Feinberg et al., 2012), at baseline, EOT and 12 months follow-up. The CRS assesses parents' perceptions of their coparenting relationship. | EOT (i.e., at 3 months postpartum) and 12 months follow-up
  The CRS consists of 35 items, divided into seven subscales that represent four theoretical coparenting domains. Total scores reflect the overall coparenting relationship, with higher scores indicating a more positive relationship. The subscale scores include agreement, closeness, support, endorsement, division, undermining, and exposure to conflict, with higher scores on the first five subscales reflecting a more positive coparenting relationship, whereas higher scores on the undermining and exposure to conflict subscales reflect a more negative coparenting dynamic.
Changes in quality of life, as measured by the EuroQol-5D-5L (EQ-5D-5L), from baseline to EOT and 12-months follow-up; | EOT (i.e., at 3 months postpartum) and 12-months follow-up
  Quality of Life as measured with the EuroQol-5D-5L (EQ-5D-5L; Herdman et al., 2011). The EQ-5D-5L measures quality of life in five dimensions of health (mobility, self-help, habitual activities, pain, anxiety/depression), each with five levels reflecting "no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems". This results in a one-digit score per dimension, which together form a five-digit code that represents the respondent's health state (e.g., 3-2-3-1-5). The sum of these digits is referred to as the severity score, indicating the overall level of reported problems. In addition, a utility index score can be calculated using a country-specific value set; in Belgium, values range from -0.532 (worst health state) to 1 (full health). The EQ Visual Analogue Scale records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labeled "the best health you can imagine" and "the worst health you can imagine".

OTHER OUTCOMES:
Cost-effectiveness, as measured by the Treatment Inventory of Costs in Patients with psychiatric disorder (TIC-P), from baseline to EOT, 6- and 12-months follow-up | EOT (i.e., at 3 months postpartum), 6- and 12-months follow-up
  Cost-effectiveness, as measured by the Treatment Inventory of Costs in Patients with psychiatric disorder (TIC-P; Bouwmans et al., 2013). The TIC-P measures medical costs and productivity losses associated with psychosocial problems in adults and is designed for use in economic evaluations. The TIC-P is a recall questionnaire, asking respondents to reflect on expenses incurred over the past one to three months.
Feasibility (1) | Baseline
  Feasibility will be investigated in terms of recruitment rate
Feasibility (2) | EOT (i.e., at 3-months post-partum)
  Feasibility will be investigated in terms of retention in treatment
Feasibility (3) | 12-months follow-up
  Feasibility will be investigated in terms of adherence to the protocol.
Acceptability (1) | EOT (i.e., at 3-months post-partum)
  Acceptability will be indicated by the number of sessions attended
Acceptability (2) | Baseline
  Acceptability will be investigated in terms of the number of individuals who refuse treatment.
Acceptability (3) | Baseline, EOT (i.e., 3-months postpartum), 12 months-follow-up
  Patient attitudes towards the treatment programs will be assessed using the Credibility and Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000) at baseline, EOT and 12 months. follow-up. The CEQ assesses patients' perceptions of how credible, logical and convincing a treatment appears, as well as their expectations regarding the improvements they believe they will achieve. The questionnaire is divided into two subscales: credibility, which reflects the perceived believability and rationality of the treatment, and expectancy, which measures the degree to which patients anticipate positive outcomes. Higher scores indicate greater treatment credibility and stronger expectations of improvement
Acceptability (4) | EOT (i.e., at months post-partum) and 12 months follow-up
  Satisfaction with treatment will be measured with the Client Satisfaction Questionnaire (CSQ; Attkinson & Greenfield 2004), at EOT and 12 months follow-up. The CSQ assesses overall participant satisfaction with an intervention. It consists of eight statements, each rated on a four-point scale. To determine the overall level of satisfaction, a total score is calculated, ranging from 8 to 32, with higher scores indicating greater satisfaction with the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luyten, PhD, Principal Investigator — University of Leuven
Locations (1):
- Obstetric outpatient clinic, UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The study results will be owned by the Sponsor. The sponsor will have access to the study data. After the publication of results focusing on primary and secondary outcomes/endpoints, anonymized data will be made available to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, ICF
Time Frame: After the publication of results focusing on primary and secondary outcomes/endpoints, anonymized data will be made available to researchers who provide a methodologically sound proposal within a reasonable time frame.